CLINICAL TRIAL: NCT01263977
Title: A Randomized Mono-center Study Looking at the Effect of Thermodilution Controlled Therapy for Volume Optimization on the Duration of Septic Shock in Patients With Septic Shock
Brief Title: Thermodilution - Controlled Management of Volume Therapy in Septic Shock
Acronym: THEMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THEMIS
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Septic Shock; Volume Status
Keywords: septic shock; goal directed volume therapy; outcome
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thermodilution controlled volume management (Experimental): Volume management based on parameters: GEDI, ELWI, CI
  Interventions: Device: Picco- thermodilution catheter
- Volume management based on surviving sepsis campaign (Active Comparator): volume management based on surviving sepsis campaign guidelines: CVP, Urin output, MAP, ScvO2
  Interventions: Device: Picco- thermodilution catheter

INTERVENTIONS:
Device: Picco- thermodilution catheter — Transpulmonary thermodilution and pulse contour analysis with arterial catheter Arterial access via femoral

SUMMARY:
Septic shock and multi-organ failure are among the most frequent causes of death in the ICU.

Patients with septic shock require early implementation of hemodynamic therapy to keep the duration of shock state and with it microcirculatory disturbances as short as possible. In the septic shock guidelines by the american association SCCM the diagnosis of volume status is based on filling pressures, like CVP. Some studies show, that the CVP depends not only on the intravascular volume, but also on the right ventricular compliance, pulmonary vascular resistance as well as intrathoracic pressure. The aim of the Study is to evaluate if the duration of septic shock can be reduced through algorithm driven volume therapy orientated to thermodilution based volume parameters (GEDI and ELWI)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from patient, authorized proxy, carer
* In women of child bearing age, effective contraceptive use with a known failure rate of <1 %
* Clinical verification of infection (≥ 48 hours possible), with at least one criteria from a - d required:

  1. Proof of pathological microorganism in blood, sputum, urine or normally sterile body tissues
  2. Identifiable focus (e.g. purulent sputum or wound secretion, perforated gut)
  3. Identification of granulocytes in normally sterile tissue
  4. Clinical suspicion of infection without identification of pathogens or micro-organisms (e.g. new pulmonary infiltrates on chest x-ray, treated pneumonia, purpura fulminants, necrotizing fasciitis)
* Confirmation of SIRS (≥ 48 hours possible), with at least 2 criteria from a-d required:

  1. Fever (≥38 °C) or Hypothermia (≤ 36 °C)
  2. Tachycardia (≥ 90/min)
  3. Tachypnoea (≥ 20/min) or Hyperventilation (PaCO2 ≤ 32 mmHg, ≤ 4,4 kPa) or mechanical ventilation
  4. Leukocytes (≥ 12,000/μl) or Leucopenia (≤ 4,000/μl) or ≥ 10% immature granulocytes
* Sepsis-induced HYPOTENSION despite adequate volume status (<24h):

Mean arterial pressure (MAP) < 65 mmHg (< 8,7 kPa) or systolic arterial pressure (SAP) < 90 mmHg (< 12 kPa) or the need for vasopressor (Norepinephrine <0.05µg/kg/min) to support the MAP ≥ 65 mmHg (≥ 8,7 kPa) or the SAP ≥ 90 mmHg ≥ 12 kPa), when one of these criteria has lasted for 4 hours or longer.

Exclusion Criteria:

* Therapy limited (DNR-Order)
* Patient moribund
* Pregnancy (positive pregnancy test in women of child bearing age)
* Breast feeding women
* Age < 18 years
* Patients active treatment for congestive heart failure with Ejection fraction < 30% and/or NYHA Class IV congestive heart failure
* Severe peripheral Arterial Vascular Occlusion Disease ≥ 2b after Fontaine
* Patients with Glasgow Coma Score ≤ 8 at the time of admission and prior to the administration of medications such as sedatives
* Patients with TNM stage 4 solid tumors, hematologic malignancies with high tumor burden, CNS tumors (WHO stage 4)
* Patients who are likely to die within days for diseases or conditions other than catecholamine-dependent shock
* Participation in another interventional clinical study within the last 30 days
* Particular relationship to senior investigator (e.g. staff, relative, colleague)
* Patients with severe liver dysfunction (Child C)
* Patients with septic shock within the last 60 days
* Patients receiving norepinephrine for longer than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Duration of septic shock | 6 months
  septic shock is defined as sepsis with mean arterial pressure (MAP) <65mmHg or systolic arterial pressure (SAP) <90mmHg or the need for vasopressors to support the MAP >/= 65 mmHg or the SAP >/= 90 mmHg

SECONDARY OUTCOMES:
28 day mortality | max 28 Tage
90 and 180 days mortality | max 180 days
Intensive care mortality | max 28 days
Frequency of arterial hypoperfusion in the extremity of the thermodilution | max. 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Claudia D Spies, MD, Prof., Study Director — Dept. of Anesthesiology and Intensive Care Medicine, CCM and CVK, Charité - Universitaetsmedizin Berlin; Michael Sander, MD, Prof., Principal Investigator — Dept. of Anesthesiology and Intensive Care Medicine, CCM and CVK, Charité - Universitaetsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte and Campus Virchow-Klinikum, Charité - Universitaetsmedizin Berlin, Berlin, State of Berlin, Germany